CLINICAL TRIAL: NCT06563804
Title: Phase 1/2 Clinical Trial of S227928, an Anti-CD74 Antibody-Drug Conjugate Targeting MCL-1, as a Single Agent and in Combination With Venetoclax in Patients With Relapsed/Refractory (R/R) Acute Myeloid Leukemia (AML), Myelodysplastic Syndrome (MDS)/AML, or Chronic Myelomonocytic Leukemia (CMML)
Brief Title: A Study to Evaluate S227928 as a Single Agent and in Combination With Venetoclax in Patients With R/R AML, MDS/AML, or CMML
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Servier Bio-Innovation LLC (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: S227928-180
Record Dates: First submitted 2024-08-14; First posted 2024-08-21 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Relapsed/Refractory (R/R) Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)/AML; Chronic Myelomonocytic Leukemia (CMML)
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation - Arm A (Experimental): S227928 as a single agent
  Interventions: Drug: S227928
- Dose Escalation - Arm B (Experimental): S227928 in combination with venetoclax
  Interventions: Drug: S227928; Drug: Venetoclax
- Dose Expansion - Cohort 1 (Experimental): For participants with R/R AML and MDS/AML. S227928 in combination with venetoclax at RP2D
  Interventions: Drug: S227928; Drug: Venetoclax
- Dose Expansion - Cohort 2 (Experimental): For participants with CMML. S227928 in combination with venetoclax at RP2D
  Interventions: Drug: S227928; Drug: Venetoclax

INTERVENTIONS:
Drug: S227928 — For administration via intravenous (IV) infusion
Drug: Venetoclax — For oral administration
  Arms: Dose Escalation - Arm B; Dose Expansion - Cohort 1; Dose Expansion - Cohort 2

SUMMARY:
The objective of this study is to determine the safety, tolerability, and anti-leukemic activity of S227928 as single agent and in combination with venetoclax, and to determine the recommended Phase 2 dose (RP2D) of this combination. The study will begin as a Phase 1 Dose Escalation study to determine the RP2D and then will transition to a Phase 2 Dose Expansion study to assess the efficacy of the selected RP2D. During the treatment period participants will have study visits every two weeks, with additional visits occurring during the first and second cycle. Approximately 30 days after treatment has ended, an end-of-treatment visit will occur and then participants will be followed for survival every 12 weeks for the next 6 months. Study visits may include a bone marrow aspirate and/or biopsy, blood and urine tests, ECG, vital signs, physical examination, and administration of study treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Women of childbearing potential (WOCBP) must use a highly effective method of birth control during study treatment and at least 6 months after the last dose of Investigational Medicinal Product (IMP). In case of the use of oral contraception, women should have been on a stable dose of the same contraceptive drug (i.e., same active principle) for at least 3 months prior to the first IMP administration.
* Male participants with WOCBP partners must use a condom during the study and for at least 3 months after the last dose of IMP. In addition, contraception should be considered for their female partners. Contraceptive measures do not apply if the participant is sterile, vasectomised or sexually abstinent. Sperm donation will not be allowed during the study and for at least 3 months after the last dose of IMP.
* Patients with pathologically confirmed AML, MDS/AML, or CMML as defined by the World Health Organization (WHO) 2022 classification or ICC, who have been previously treated with at least one prior standard treatment and have relapsed and/or refractory disease.

  1. Patients must not be candidates for further standard therapy,
  2. Treatment with agents for lower risk MDS such as erythropoietin or luspatercept are not considered anticancer therapies.
* Circulating leukocytes < 10 x 109/L (use of hydroxycarbamide before study drug initiation is allowed to achieve this inclusion criterion).
* Adequate renal function within 7 days before study enrollment defined as:

  a. Calculated creatinine clearance (determined by the modification of diet in renal disease [MDRD] equation) ≥ 60 mL/min
* Adequate hepatic function within 7 days before study enrollment defined as:

  1. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN),
  2. Total bilirubin level ≤ 1.5 x ULN, except for patients with known Gilbert's syndrome, who may be included if their total bilirubin is ≤ 3.0 x ULN and their direct bilirubin is ≤ 1.5 x ULN.

Key Exclusion Criteria:

* Pregnant or lactating women.
* WOCBP tested positive in a serum pregnancy test within 7 days prior to the first day of IMP administration.
* Legally incapacitated person under guardianship or trusteeship.
* Failure to recover to ≤ Grade 1 (Common Terminology Criteria for Adverse Events version 5.0 [CTCAE v5.0]) from acute non-hematologic toxicities (to ≤ Grade 2 for neuropathy) due to previous therapy, prior to screening.
* Diagnosis of myeloproliferative neoplasms (MPNs) or other non-CMML MDS/MPNs as defined by the WHO 2022 classification
* Diagnosis of acute promyelocytic leukemia (French-American-British [FAB] M3 classification).
* Diagnosis of acute leukemia of mixed or ambiguous lineage or histiocytic/dendritic cell neoplasms defined by the WHO 2022 classification
* Uncontrolled infections requiring systemic antibiotics and/or antifungal agents as per investigator's judgment. Patients receiving prophylactic antibiotics and/or antifungal agents are eligible for this study.
* Serologic evidence of chronic hepatitis B virus (HBV) infection and unable or unwilling to receive standard prophylactic antiviral therapy, or with detectable HBV viral load.
* Serologic evidence of hepatitis C virus (HCV) infection without completion of curative treatment or with detectable HCV viral load.
* Human immunodeficiency virus (HIV) seropositive with any of the following:

  1. CD4+ T-cell (CD4+) counts < 350 cells/µL
  2. Acquired immunodeficiency syndrome-defining opportunistic infection within 12 months prior to screening
  3. Not on antiretroviral therapy, or on antiretroviral therapy for < 6 weeks at the time of Day 1 in Cycle 1
  4. HIV viral load ≥ 400 copies/mL
* Participants with a known clinically significant cardiovascular disease or condition, including

  1. Uncontrolled arterial hypertension per the investigator's judgment
  2. New York Heart Association class III or IV congestive heart failure
  3. Congenital or substance-induced long QT defined as heart rate-corrected QT (QTc) interval >450 ms for males and >470 ms for females according to Fridericia's formula
  4. Uncontrolled cardiac arrhythmia (e.g., participants with rate-controlled atrial fibrillation are eligible)
  5. Severe uncorrected conduction disturbances (e.g., 3rd degree heart block). Patients with severe conduction disturbances corrected by a pacemaker are eligible
  6. Acute coronary syndrome (including unstable angina pectoris, acute myocardial infarction), coronary angioplasty or bypass grafting within 6 months prior to the first IMP administration
  7. Troponin I > ULN or troponin T > ULN if troponin I cannot be assessed
  8. Any factors that could increase the risk of QTc interval prolongation or risk of arrhythmic events such as heart failure, family history of QT syndrome, or family history of unexplained sudden death under 40 years of age
* Known active central nervous system involvement by AML, MDS/AML, or CMML.
* Coagulation disorders or abnormalities that may increase the risk of bleeding complications according to investigator's judgment (e.g., disseminated intravascular coagulation).
* Any clinically significant medical condition (e.g., organ dysfunction, gastric ulcer) or laboratory abnormality likely to jeopardize the patient's safety or to interfere with the conduct of the study.
* Major surgery within 4 weeks before the first IMP administration, or patients who have not recovered from the acute effects of surgery.
* Allogeneic stem cell transplantation (SCT) within 3 months before the first dose of IMP

  a. Patients cannot be receiving any immunosuppressive treatment, except for corticosteroids used as physiologic replacement doses up to the equivalent of 10 mg of oral prednisone
* Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: 1) malignancies that were treated curatively, which have not recurred within 3 years prior to study entry and do not require further treatment; 2) completely resected basal and squamous cell skin cancers; 3) any malignancy considered to be indolent and that has never required anticancer therapy; and 4) completely resected carcinoma in situ of any type.
* History of severe allergic or anaphylactic reactions to BH3 mimetics (including venetoclax) or to any excipients of S227928.
* Any previous anticancer treatment for the studied disease within 2 weeks or at least 5 half-lives (whichever is longer) prior to first dose of IMPs (except for hydroxycarbamide). In case of investigational biologic agents with a long half-life, such as immune checkpoint or bispecific antibodies, a flat wash-out period of 28 days will be acceptable. Participation in non-interventional registries or epidemiological studies is allowed. Hormonal therapies are not considered anticancer treatments for eligibility purposes.
* Any cellular therapies (e.g., NK or CAR T cells) within 100 days prior to first dose of IMP.
* Any radiotherapy within 2 weeks before the first dose of IMPs (except for palliative radiotherapy to localized lesions, i.e., chloromas).
* Any drugs known to prolong the QT interval and induce Torsade de pointes (TdP) within 7 days prior to the first administration of IMP.
* Dose Escalation Arm A ONLY: Although participants may be treated with strong inhibitors of CYP3A4 or of CYP2C8, they may not be treated with medications that are strong inhibitors of both CYP3A4 and CYP2C8, or with separate medications that when combined would cause strong inhibition of these two enzymes. In addition, participants may not be treated with a strong inhibitor of CYP3A4 and a moderate inhibitor of CYP2C8 and/or a moderate inhibitor of P-gp. These prohibitions begin 7 days prior to the start of IMP and continue for the entire duration of treatment. Triazole antifungal agents may be used, but only if they are in agreement with the criteria described above (i.e., they must not be dual strong inhibitors of both CYP3A4 and CYP2C8 or strong inhibitors of CYP3A4 and moderate inhibitors of either CYP2C8 or P-gp).
* Dose Escalation Arm B and Dose Expansion ONLY: a malabsorption syndrome or other condition that precludes enteral route of administration.
* Dose Escalation Arm B and Dose Expansion ONLY: Both moderate and strong inhibitors of CYP3A4 are prohibited, beginning 7 days prior to the start of IMP and continuing for the entire duration of treatment.
* Dose Escalation Arm B and Dose Expansion ONLY: Both moderate and strong CYP3A4 inducers are prohibited, beginning 14 days before the start of IMP and continuing for the entire duration of treatment.
* Dose Escalation Arm B and Dose Expansion ONLY: treatment with P-gp and BCRP inhibitors; or with medications with a narrow therapeutic index (NTIs) which are substrates of P-gp or BCRP; or with OATP1B1 substrates that cannot be discontinued 7 days before and during study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Number and severity of Dose Limiting Toxicities (DLTs) | Through Cycle 1 (each cycle is 28 days)
Dose Escalation: Number of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Through 30 days after the end of treatment (Approximately 3.5 years)
Dose Escalation: Number of dose reductions, interruptions, delays, or study withdrawal due to AEs | Through 30 days after the end of treatment (Approximately 3.5 years)
Dose Expansion: Complete remission (CR) | Through 6 months after the end of treatment (Approximately 4 years)

SECONDARY OUTCOMES:
Dose Escalation: Cmax of S227928, total Monoclonal Antibody (mAb), and unconjugated S64315 | Through the end of treatment (Approximately 3.5 years)
Dose Expansion: Cmax of S227928, total mAb, and unconjugated S64315 | Through the end of treatment (Approximately 3.5 years)
Dose Escalation: Tmax of S227928, total mAb, and unconjugated S64315 | Through the end of treatment (Approximately 3.5 years)
Dose Expansion: Tmax of S227928, total mAb, and unconjugated S64315 | Through the end of treatment (Approximately 3.5 years)
Dose Escalation: Area Under the Curve (AUC) of S227928, total mAb, and unconjugated S64315 | Through the end of treatment (Approximately 3.5 years)
Dose Expansion: AUC of S227928, total mAb, and unconjugated S64315 | Through the end of treatment (Approximately 3.5 years)
Dose Escalation: Plasma concentration vs. time profile of S227928 | Through the end of treatment (Approximately 3.5 years)
Dose Expansion: Plasma concentration vs. time profile of S227928 | Through the end of treatment (Approximately 3.5 years)
Dose Escalation: Plasma concentration vs. time profile of unconjugated S64315 | Through the end of treatment (Approximately 3.5 years)
Dose Expansion: Plasma concentration vs. time profile of unconjugated S64315 | Through the end of treatment (Approximately 3.5 years)
Dose Escalation: Plasma concentration vs. time profile of total mAb | Through the end of treatment (Approximately 3.5 years)
Dose Expansion: Plasma concentration vs. time profile of total mAb | Through the end of treatment (Approximately 3.5 years)
Dose Escalation (Arm B ONLY): Plasma concentration vs. time profile of venetoclax | Through the end of treatment (Approximately 3.5 years)
Dose Expansion: Plasma concentration vs. time profile of venetoclax | Through the end of treatment (Approximately 3.5 years)
Dose Escalation: Detection of Anti-Drug Antibodies (ADAs) against S227928 | Through the end of treatment (Approximately 3.5 years)
Dose Expansion: Detection of ADAs against S227928 | Through the end of treatment (Approximately 3.5 years)
Dose Escalation: Complete remission (CR) | Through 6 months after the end of treatment (Approximately 4 years)
  For patients with R/R AML or MDS/AML, or R/R CMML
Dose Escalation: Complete remission with incomplete hematologic recovery (CRi) | Through 6 months after the end of treatment (Approximately 4 years)
  For patients with R/R AML or MDS/AML
Dose Expansion: CRi | Through 6 months after the end of treatment (Approximately 4 years)
  Cohort 1 only
Dose Escalation: Morphologic leukemia-free state (MLFS) | Through 6 months after the end of treatment (Approximately 4 years)
  For patients with R/R AML or MDS/AML
Dose Expansion: MLFS | Through 6 months after the end of treatment (Approximately 4 years)
  Cohort 1 only
Dose Escalation: CR with partial hematologic recovery (CRh) | Through 6 months after the end of treatment (Approximately 4 years)
  For patients with R/R AML or MDS/AML, or R/R CMML
Dose Expansion: CRh | Through 6 months after the end of treatment (Approximately 4 years)
Dose Escalation: Partial remission (PR) | Through 6 months after the end of treatment (Approximately 4 years)
  For patients with R/R AML or MDS/AML, or R/R CMML
Dose Expansion: PR | Through 6 months after the end of treatment (Approximately 4 years)
Dose Escalation: Overall survival (OS) | Through 6 months after the end of treatment (Approximately 4 years)
  For patients with R/R AML or MDS/AML, or R/R CMML
Dose Expansion: OS | Through 6 months after the end of treatment (Approximately 4 years)
Dose Escalation: Duration of response (DOR) | Through 6 months after the end of treatment (Approximately 4 years)
  For patients with R/R AML or MDS/AML
Dose Expansion: DOR | Through 6 months after the end of treatment (Approximately 4 years)
  Cohort 1 only
Dose Escalation: Time to first remission (CR or CRh or CRi) | Through 6 months after the end of treatment (Approximately 4 years)
  For patients with R/R AML or MDS/AML
Dose Expansion: Time to first remission (CR or CRh or CRi) | Through 6 months after the end of treatment (Approximately 4 years)
  Cohort 1 only
Dose Escalation: Red-blood cell (RBC) and platelet transfusion independence for at least 8 weeks | Through 6 months after the end of treatment (Approximately 4 years)
  For patients with R/R AML or MDS/AML
Dose Expansion: RBC and platelet transfusion independence for at least 8 weeks | Through 6 months after the end of treatment (Approximately 4 years)
  Cohort 1 only
Dose Escalation: CR with limited count recovery (CRL) | Through 6 months after the end of treatment (Approximately 4 years)
  For patients with R/R CMML
Dose Expansion: CRL | Through 6 months after the end of treatment (Approximately 4 years)
  Cohort 2 only
Dose Escalation: CR equivalent | Through 6 months after the end of treatment (Approximately 4 years)
  For patients with R/R CMML
Dose Expansion: CR equivalent | Through 6 months after the end of treatment (Approximately 4 years)
  Cohort 2 only
Dose Escalation: Hematologic improvement (HI) | Through 6 months after the end of treatment (Approximately 4 years)
  For patients with R/R CMML
Dose Expansion: HI | Through 6 months after the end of treatment (Approximately 4 years)
  Cohort 2 only
Dose Escalation: Overall response rate (ORR)= CR + CR equivalent + CRh + CRL + PR + HI | Through 6 months after the end of treatment (Approximately 4 years)
  For patients with R/R CMML
Dose Expansion: Overall response rate (ORR)= CR + CR equivalent + CRh + CRL + PR + HI | Through 6 months after the end of treatment (Approximately 4 years)
  Cohort 2 only
Dose Escalation: Progression-free survival (PFS) | Through 6 months after the end of treatment (Approximately 4 years)
  For patients with R/R CMML
Dose Expansion: PFS | Through 6 months after the end of treatment (Approximately 4 years)
  Cohort 2 only
Dose Escalation: Event-free survival (EFS) | Through 6 months after the end of treatment (Approximately 4 years)
  For patients with R/R CMML
Dose Expansion: EFS | Through 6 months after the end of treatment (Approximately 4 years)
Dose Expansion: Number and severity of Dose Limiting Toxicities (DLTs) of S227928 in combination with venetoclax | Through Cycle 1 (each cycle is 28 days)
Dose Expansion: AEs and SAEs | Through 30 days after the end of treatment (Approximately 3.5 years)
Dose Expansion: Number of dose reductions, interruptions, delays, or study withdrawal due to AEs | Through 30 days after the end of treatment (Approximately 3.5 years)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (5):
  - City of Hope, Duarte, California
  - The University of Kansas, Fairway, Kansas
  - START Midwest, Grand Rapids, Michigan
  - Memorial Sloan Kettering, New York, New York
  - Fred Hutch Cancer Center, Seattle, Washington
- Australia (2):
  - Peter MacCallum Cancer Centre, Melbourne
  - Prince of Wales Hospital, Randwick
- Helsinki University Hospital - Comprehensive Cancer Center, Helsinki, Finland
- France (4):
  - Institut Paoli Calmette, Marseille
  - Chu de Nice - Hôpital L'archet 1, Nice
  - CHU de Bordeaux - Hopital du Haut Levêque, Pessac
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Klinikum rechts der Isar der TU München, München
  - Universitätsklinikum Ulm, Ulm
- Japan (2):
  - Sapporo Hokuyu Hospital, Hokkaido
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data. Access can be requested for all interventional clinical studies:
  * Used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * Sponsored by Servier
  * With a first patient enrolled as of 1 January 2004 onwards
  * For New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/